CLINICAL TRIAL: NCT01065233
Title: Genetical Predisposition in Hepatocellular Carcinoma : Pangenomic Link Study During Alcoholic Cirrhosis
Brief Title: Pangenomic Study During Alcoholic Cirrhosis
Acronym: CDCHC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/07/08-M
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Alcoholic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 blood samples of 5ml for DNA extraction

GROUPS / COHORTS (2):
- alcoholic cirrhosis with viral infection: patient with alcoholic cirrhosis with viral infection (300 patients)
  Interventions: Genetic: DNA extraction
- alcoholic cirrhosis without viral infection: patient with alcoholic cirrhosis without viral infection
  Interventions: Genetic: DNA extraction

INTERVENTIONS:
Genetic: DNA extraction — DNA extraction of blood sample for DNAship analysis

SUMMARY:
Hepatocellular carcinoma (HCC) is a frequent complication of cirrhosis. Occurrence of HCC could be linked with multiple functional region of genome.

The determining of a genomic mapping of " single nucleotide polymorphisms " (SNPs) permit to perform some genetic link studies with pathologies without clear hereditary disposition.

In this study, the investigators will identify predictives genetic polymorphism of HCC.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 70 years old
* Compensated cirrhosis or not
* Caucasian origin of the parents
* Patient with cirrhosis (histological proof or obvious)

Exclusion Criteria:

* HIV, HBV, HCV positive
* Known Homozygotia (C282Y+/+)
* Important hepatocytary iron overload for patient with resection
* HCC non histologically prooved

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2 groups with 2 subgroups:
  * patient with HCC
  * HCC with Child A
  * HCC with Child B/C
  * patient without HCC
  * Child A without HCC
  * Child B/C without HCC
Sampling Method: Probability Sample
Enrollment: 1325 (Actual)
Dates: Start 2008-10-23 (Actual); Primary Completion 2011-12-27 (Actual); Study Completion 2013-07-20 (Actual)

PRIMARY OUTCOMES:
Existence of HCC and Pangenomic analysis of DNA polymorphism
  Existence of HCC and determination of which genetic polymorphism are predisposing to HCC or preventing for HCC

SECONDARY OUTCOMES:
cirrhosis severity (compensated or not)
  Analysis of the genetic polymorphism involved in the severity of cirrhosis

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Nantes UH, Nantes
  - Jean Verdier UH, Paris
  - Paul Brousse UH, Paris
  - Rennes UH, Rennes

REFERENCES:
- [Derived] Archambeaud I, Auble H, Nahon P, Planche L, Fallot G, Faroux R, Gournay J, Samuel D, Kury S, Feray C. Risk factors for hepatocellular carcinoma in Caucasian patients with non-viral cirrhosis: the importance of prior obesity. Liver Int. 2015 Jul;35(7):1872-6. doi: 10.1111/liv.12767. Epub 2015 Jan 21. PMID 25522809